CLINICAL TRIAL: NCT04757857
Title: Randomized, Pragmatic, Open Controlled Multicentre Study, Evaluating the Use of Rivaroxaban in Mild or Moderate COVID-19 Patients
Brief Title: COVID-19 Antithrombotic Rivaroxaban Evaluation
Acronym: CARE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sustained reduction in the number of new COVID-19 cases as well as lower than expected event rates
Sponsor: Hospital Alemão Oswaldo Cruz (Other)
Collaborators: Bayer (Industry); Hospital Israelita Albert Einstein (Other); Hospital do Coracao (Other); Hospital Sirio-Libanes (Other); Hospital Moinhos de Vento (Other); Brazilian Research In Intensive Care Network (Network); Brazilian Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Álvaro Avezum Junior, Research Manager - International Research Center, Hospital Alemão Oswaldo Cruz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36066320.5.1001.0070
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: SARS-Cov-2; COVID-19; Rivaroxaban; Antithrombotic
MeSH Terms: conditions — COVID-19 | interventions — Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Pragmatic, open-label, controlled randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban 10 mg (Active Comparator): Participants will receive, from the 1st to the 14th day, a dose of 10 mg of rivaroxaban - OA (Oral Administration).
  Interventions: Drug: Rivaroxaban 10 mg
- Best locally standardized care (No Intervention): According to the study protocol, participating investigators are advised to follow the best available local practice in each participating site. There is no formal recommendation for any particular COVID-19 treatment, except symptomatic therapies.

INTERVENTIONS:
Drug: Rivaroxaban 10 mg — Rivaroxaban pharmaceutical form will be tablets of 10 mg
  Other Names: Xarelto
  Arms: Rivaroxaban 10 mg

SUMMARY:
There are several ways in which the COVID-19 pandemic may affect the prevention and management of thrombotic and thromboembolic disease, either direct effect or the indirect effects of infection, such as through severe illness and hypoxia, may predispose patients to thrombotic events. The severe inflammatory response, critical illness, and underlying traditional risk factors may all predispose to thrombotic events. Therefore, considering the high-risk profile of cardiovascular comorbidities in patients with COVID-19, it is scientifically relevant to evaluate the use of anticoagulants as an adjunctive treatment in the context of COVID-19. Indeed, it will be tested the hypothesis that the use of moderate dose of rivaroxaban has a beneficial effect in the treatment of patients with a confirmed or probable diagnosis of COVID-19 infection, with no clear indication for hospitalization (mild and moderate cases) upon initial medical care, by reducing the need of hospitalization due to complications related to COVID-19.

DETAILED DESCRIPTION:
Initial studies suggest an inflammatory state and hypercoagulation in individuals with COVID-19. Apparently, the fact that the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) spike protein binds to Angiotensin Converting Enzyme 2 (ACE2) receptors can lead to ACE2 depletion by SARS-CoV-2 favoring the "harmful" ACE1 / angiotensin II and promoting tissue damage, including stroke. Recent observational studies indicate a higher rate of thromboembolism in patients with COVID-19, especially those in severe condition. They also report that, in patients treated with anticoagulants, complication rates were lower as compared with those not receiving anticoagulant therapies.

More recently, in a post-mortem study of patients with Covid-19 compared to recently published cases of influenza, the histopathological pattern on the periphery of the lungs of patients with Covid-19 revealed a diffuse alveolar lesion with infiltration of perivascular T cells and other vascular aspects, consisting of severe endothelial damage (endothelitis) associated with the presence of intracellular viruses and broken cell membranes. In addition, pulmonary vessels showed generalized thrombosis with microangiopathy, and alveolar capillary microthrombi were much more frequent in patients with COVID-19 than with severe influenza respiratory conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years old;
2. Evaluated in the emergency unit with probable or confirmed infection by COVID-19;
3. Time between symptoms and inclusion ≤ 07 days *;
4. Present mild or moderate signs and symptoms, with no clear indication for hospitalization;
5. Present at least 2 risk factors for complication:

   * 65 years
   * Hypertension
   * Diabetes mellitus
   * Asthma
   * Chronic Obstructive Pulmonary Disease (COPD) or other chronic lung diseases
   * Smoking
   * Immunosuppression
   * Obesity (BMI> 30)
   * History of non-active cancer
   * Bed restriction or reduced mobility (≥50% of the wake time without walking)
   * Previous history of VTE
   * Use of oral hormonal contraceptives

Exclusion Criteria:

1. Patients <18 years old;
2. Hospitalization indication upon first medical care;
3. Positive test for influenza in the first visit;
4. Any known liver disease associated with coagulopathy; INR (International Normalized Ratio) > 1.5;
5. Pregnant, lactating or with the possibility of becoming pregnant and without using an adequate contraceptive method;
6. High risk of bleeding; History of bronchiectasis or pulmonary cavitation, Significant bleeding in the last 3 months, Active gastroduodenal ulcer, history of recent bleeding (within 3 months) or a high risk of bleeding;
7. Stroke within 1 month or any history of hemorrhagic or lacunar stroke or any intracranial bleeding or any intracranial neoplasia, brain metastasis, arteriovenous malformation or brain aneurysm;
8. Severe heart failure with left ventricular ejection fraction <30% (echocardiogram or other validated method previously documented) or symptoms of heart failure class III or IV of the New York Heart Association (NYHA);
9. Estimated glomerular filtration rate (eGFR) <30 mL / min;
10. Clinical indication for dual antiplatelet therapy or anticoagulation therapy (VTE, atrial fibrillation / flutter, mechanical valve prosthesis);
11. Marked thrombocytopenia (platelets <50,000 / mm3);
12. Non-cardiovascular disease that is associated with a poor prognosis, for example, active cancer (excluding non-melanoma skin cancer) defined as cancer without remission or requiring active chemotherapy or adjuvant therapies such as immunotherapy or radiation therapy or that increases the risk of an adverse reaction to the evaluated interventions;
13. History of hypersensitivity or known contraindication to rivaroxaban;
14. Systemic treatment with strong inhibitors of Cytochrome P450 3A4 (CYP3A4) and glycoprotein p (Pgp) (for example, systemic azole antimycotics, such as ketoconazole and human immunodeficiency virus [HIV] protein inhibitors, such as ritonavir) or strong inducers of CYP 3A4, that is, rifampicin, rifabutin, phenobarbital, phenytoin and carbamazepine;
15. Current treatment being tested;
16. Concomitant participation in another study with experimental drugs in the context of COVID;
17. Use of chloroquine or hydroxychloroquine associated with azithromycin;
18. Active cancer;
19. Other contraindications to rivaroxaban;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolic events (VTE) | Within 30 days from randomization
  Defined as deep venous thrombosis, acute pulmonary embolism, other major venous thrombotic events.
Mechanical ventilation free-survival | Within 30 days from randomization
  Defined as survival without requirement of mechanical ventilation.
Major Adverse Cardiovascular Events (MACE) | Within 30 days from randomization
  Defined as acute myocardial infarction, stroke or acute limb ischemia
Out-of-hospital death not attributed to major injury | Within 30 days from randomization
  Death that occurred out of hospital due to any cause not related to trauma or other major injury

SECONDARY OUTCOMES:
Time from randomization to hospitalization | 30 days from randomization
  Defined as time elapsed since randomization to hospital admission
Length of Hospitalization | 30 days from randomization
  To assess the duration of hospitalization (length of hospital stay)
Hospitalization in Intensive Care Unit | 30 days from randomization
  Requirement of admission to ICU for intensive care
Clinical requirement of mechanical ventilation | 30 days from randomization
  Requirement of oxygen supplementation through invasive or non invasive mechanical ventilation.
Clinical duration of mechanical ventilation | 30 days from randomization
  Total time on oxygen supplementation through invasive or non invasive mechanical ventilation
Composite vascular endpoint I | 30 days from randomization
  Non-fatal myocardial infarction, non-fatal ischemic stroke or cardiovascular death, VTE
Composite vascular endpoint II | 30 days from randomization
  Cardiovascular death, non-fatal myocardial infarction, non-fatal ischemic stroke or acute limb ischemia, VTE
Major Bleeding | 30 days from randomization
  Defined by International Society of Thrombosis and Hemostasis (ISTH) criteria
Mortality | 30 days from randomization
  Defined by all-cause deaths

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro Avezum, Ph.D, Principal Investigator — International Research Center - Hospital Alemão Oswaldo Cruz
Locations (36):
- Brazil (36):
  - Hospital Maternidade São Vicente de Paulo, Barbalha, Ceará
  - Clínica Senhor do Bonfim, Feira de Santana, Estado de Bahia
  - Hospital de Base do Distrito Federal, Brasília, Federal District
  - Hospital de Campanha Covid-19 Goiânia/Sesgo, Goiânia, Goiás
  - Hospital Estadual de Urgências de Trindade/SESGO, Trindade, Goiás
  - Núcleo de Pesquisa Clínica do Hospital Vera Cruz, Belo Horizonte, Minas Gerais
  - Hospital São Lucas, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericórdia de Passos, Passos, Minas Gerais
  - Hospital Universitário Regional de Maringá, Maringá, Paraná
  - Beneficencia Nipo Brasileira Da Amazonia, Belém, Pará
  - Hospital Adventista de Belém, Belém, Pará
  - Associação Dr. Bartholomeu Tacchini, Bento Gonçalves, Rio Grande do Sul
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital das Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Universitario de Santa Maria, Santa Maria, Rio Grande do Sul
  - Clínica Procárdio Ltda, Blumenau, Santa Catarina
  - H&W Cardiologia LTDA, Joinville, Santa Catarina
  - Irmandade santa Casa de Araras, Araras, São Paulo
  - Alphacor Cardiologia Clínica e Diagnóstica LTDA, Barueri, São Paulo
  - Maestri e Kormann Consultoria Medico-Cientifica LTDA - EPP, Blumenau, São Paulo
  - Hospital Regional do Litoral Norte - Instituto Sócrates Guanaes, Caraguatatuba, São Paulo
  - Hospital Santos Dumont Litoral Norte, Caraguatatuba, São Paulo
  - Hospital de Corderiopolis, Cordeirópolis, São Paulo
  - Hospital Regional Jorge Rossman - Instituto Sócrates Guanaes, Itanhaém, São Paulo
  - Hospital Carlos Fernando Malzoni, Matão, São Paulo
  - Hospital Moinhos de Vento, Porto Alegre, São Paulo
  - Hospital Regional de Registro - Instituto Sócrates Guanaes, Registro, São Paulo
  - Hospital Unimed Ribeirão Preto, Ribeirão Preto, São Paulo
  - Kaiser Clinica e Hospital Dia, São José do Rio Preto, São Paulo
  - Braile Hospital Dia Ltda, São José do Rio Preto, São Paulo
  - Hospital Policlin, São José dos Campos, São Paulo
  - Hospital Regional de São José dos Campos - Instituto Sócrates Guanaes, São José dos Campos, São Paulo
  - Santa Casa de Misericórdia de Votuporanga, Votuporanga, São Paulo
  - International Research Center - Hospital Alemão Oswaldo Cruz, São Paulo
  - Hospital Leforte Liberdade, São Paulo
  - Incor - Instituto do Coração do Hospital das Clínicas da FMUSP, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santos BC, Flumignan RL, Civile VT, Atallah AN, Nakano LC. Prophylactic anticoagulants for non-hospitalised people with COVID-19. Cochrane Database Syst Rev. 2023 Aug 16;8(8):CD015102. doi: 10.1002/14651858.CD015102.pub2. PMID 37591523
- [Derived] Avezum A, Oliveira Junior HA, Neves PDMM, Alves LBO, Cavalcanti AB, Rosa RG, Veiga VC, Azevedo LCP, Zimmermann SL, Silvestre OM, Seabra Prudente RC, Morales Kormann AP, Moreira FR, Boszczowski I, de Brito Sobrinho E, da Silva E Souza A, Seligman R, de Souza Paolino B, Razuk A, Diogenes de Magalhaes Feitosa A, Monteiro Belmonte PL, Freitas das Neves Goncalves P, Hernandes ME, Fagundes AL, Sarmet Esteves JM, Tognon AP, Eikelboom J, Berwanger O, Lopes RD, Oliveira GBF; Coalition VIII COVID-19 Brazil Investigators. Rivaroxaban to prevent major clinical outcomes in non-hospitalised patients with COVID-19: the CARE - COALITION VIII randomised clinical trial. EClinicalMedicine. 2023 Jun;60:102004. doi: 10.1016/j.eclinm.2023.102004. Epub 2023 May 18. PMID 37223666
- [Derived] Oliveira GBF, Neves PDMM, Oliveira HA, Catarino DGM, Alves LBO, Cavalcanti AB, Rosa RG, Veiga VC, Azevedo LCP, Berwanger O, Lopes RD, Avezum A. Rivaroxaban in Outpatients with Mild or Moderate COVID-19: Rationale and Design of the Study CARE (CARE - Coalition COVID-19 Brazil VIII). Arq Bras Cardiol. 2023 Mar;120(3):e20220431. doi: 10.36660/abc.20220431. English, Portuguese. PMID 37018790